CLINICAL TRIAL: NCT00322816
Title: Malaria Prevalence, Incidence and Mortality in Children
Brief Title: Malaria Prevalence in Children
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: 05-0068
Record Dates: First submitted 2006-05-04; First posted 2006-05-08 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2011-11

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Malaria, Plasmodium falciparum, Gambia, larvicides
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this pilot study is to evaluate the use of (1) 'malaria prevalence', (2) 'malaria incidence' and (3) 'malaria mortality' as a measure of malaria transmission in The Gambia, while mosquito insecticides (larvicides) are used to control malaria-carrying mosquitoes. Two thousand children aged 6 months to 10 years of age will be recruited from villages in the study area. They will be monitored over 7 months for the presence of malaria parasites and signs and symptoms of the disease.

DETAILED DESCRIPTION:
Malaria remains one of the world's greatest childhood killers and is a substantial obstacle to social and economic development in the tropics. The overwhelming bulk of the world's malaria burden rests upon the population of sub-Saharan Africa because of the unique coincidence of expanding human populations, weak health systems, the world's most effective vector mosquito species and environmental conditions ideal for transmission. At the start of the new millennium malaria is still deeply entrenched in Africa and effective malaria control is under threat from the inexorable spread of parasite strains resistant to antimalarial drugs and the emergence of mosquitoes resistant to the pyrethroid insecticides used to impregnate bednets. Larval control may offer a new alternative for effective control. We plan to apply a larvicide in an effort to control malaria and reduce the burden of malaria. While it is abundantly clear that this product will kill mosquito larvae in the laboratory and in the field, it is not certain that doing so will reduce the burden of malaria for the human population. There are several steps which intervene between the survival of mosquito larvae in aquatic breeding sites and the human end points that we hope to achieve. Briefly, the steps involved include survival and development of immature mosquito stages, emergence of adult mosquitoes, blood feeding by those mosquitoes, acquisition and development of malaria parasites by adult mosquitoes and transmission of parasites to susceptible humans. Once infected, the human population may either clear the infection over time or go on to develop symptoms. Among those who develop symptoms, some receive prompt and successful treatment, while some others go on to either develop chronic symptoms or to progress through severe malaria to death. Primary outcomes are: 1) the proportion of subjects with malaria parasites (Plasmodium Falciparum), 2) the incidence of clinical malaria, and 3) the age-standardized overall and malaria-specific mortality. Secondary outcomes are: 1) prevalence of a clinical episode of malaria (presence of malaria parasites plus an axillary temperature of 37.5 C or greater during examination or a history of fever during the last 48 hours); 2) prevalence of high parasitemias (defined as equal to of greater than 5000 parasites per mcl); 3) prevalence of enlarged spleen (defined using Hackett's classification); and 4) prevalence of severe anemia (defined as hemoglobin less than or equal to 5 g/dl). Within a broad area of eastern Gambia, zones have been identified for application of larvicide, with matched control zones where no larval control have been applied. In each area, the human population will be monitored to determine whether one of four specific malariometric end points will provide a valid assessment of larvicidal effectiveness. In this study 2000 children, 6 months to 10 years of age, will be recruited. These pilot studies will inform subsequent (not included in this NIH project) large scale evaluations of larviciding for malaria control. This protocol is designed to determine whether prevalence and incidence of malaria attacks and deaths can be used to evaluate the impact of Bti for malaria transmission control.

ELIGIBILITY:
Inclusion Criteria:

All children living in the defined areas for intervention and between the age of 6 months and 10 years will be invited to participate. No distinctions will be made regarding gender or ethnic group. Moreover, as the target population is all people living in the areas of intervention, and in order of the results from this study to be as generalizable as possible, no distinctions will be made in terms of medical condition or physical health. Moreover, we believe that any children with a medical condition would be especially favored by the participation in the study.

Exclusion Criteria:

None

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2552 (Actual)
Dates: Start 2006-06-07; Primary Completion 2008-03-31 (Actual); Study Completion 2009-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Council's Laboratories, Fajara, The Gambia